CLINICAL TRIAL: NCT00669071
Title: Split-Face, Randomized, Open-Label Study of Sequential Treatment With Tri-Luma® Cream With Intense Pulsed Light (IPL) vs. a Mild Inactive Control Cream With Intense Pulsed Light (IPL) in Subjects With Melasma
Brief Title: Treatment w/ Tri-Luma® Cream & Intense Pulsed Light (IPL) vs a Mild Inactive Control Cream & Intense Pulsed Light (IPL) in Melasma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment closed
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: US10081
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2012-09

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Fluocinolone Acetonide; hydroquinone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPL / Tri-Luma® Cream (Active Comparator)
  Interventions: Drug: Fluocinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05%
- IPL/Cetaphil® Moisturizing Cream as Inactive Control (Active Comparator)
  Interventions: Drug: Cetaphil® Moisturizing Cream as Inactive Control

INTERVENTIONS:
Drug: Fluocinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05% — Applied once daily at bedtime on one side of the face; this was a randomized, split face study where one cream was used on the right side of the face and the other cream on the left side of the face and IPL (Intense Pulsed Light) was used on both sides of the face.
  Other Names: Tri-Luma® Cream
  Arms: IPL / Tri-Luma® Cream
Drug: Cetaphil® Moisturizing Cream as Inactive Control — Applied once daily at bedtime on the opposite side of the face; this was a randomized, split face study where one cream was used on the right side of the face and the other cream on the left side of the face and IPL (Intense Pulsed Light) was used on both sides of the face.
  Other Names: Cetaphil® Moisturizing Cream
  Arms: IPL/Cetaphil® Moisturizing Cream as Inactive Control

SUMMARY:
This study is to evaluate the efficacy and safety of Tri-Luma® Cream (fluocinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05%) when used sequentially with a series of intense pulsed light (IPL) treatments in Subjects diagnosed with moderate to severe melasma during a 10 week treatment period.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with moderate to severe melasma on both sides of the face (Investigator's Global Assessment (IGA) at baseline must be 3 or 4.)

Exclusion Criteria:

* Subjects with a diagnosis of skin cancer (Basal Cell Carcinoma (BCC), Squamous Cell Carcinoma (SCC), Melanoma) in the areas to be treated
* Subjects with prior facial Intense Pulsed Light (IPL), resurfacing, deep or chemical peels within 6 months of the date of study entry
* Subject has initiated treatment with hormones including estrogen, progesterone and/or oral contraceptives within 3 months of study entry, or who intend to discontinue hormonal therapy during the study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron W Gottschalk, MD, Study Director — Galderma R&D
Locations (2):
- United States (2):
  - Dermatology/Cosmetic Laser Associates of La Jolla, Inc., La Jolla, California
  - Tennessee Clinical Research Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on January 8, 2008 and the last subject was enrolled on August 6, 2008.
Pre-assignment Details: The specified wash-out period up to baseline was:
  * 2 weeks since the use of Non-Steroidal Anti- Inflammatory Drugs (NSAIDs)
  * 14 days for melasma treatments at the time of study entry or under current treatment
  * at least 6 months since prior facial IPL, resurfacing, deep or chemical peels from the date of study entry
Groups:
- IPL / Tri-Luma® Cream and IPL / Inactive Control Cream: Intense Pulsed Light (IPL)/fluocinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05% cream (Tri-Luma® Cream) and Intense Pulsed Light (IPL)/Cetaphil® Moisturizing Cream; Applied once daily at bedtime on one side of the face; this was a randomized, split face study where one cream was used on the right side of the face and the other cream on the left side of the face and IPL (Intense Pulsed Light) was used on both sides of the face.
Period: Overall Study
Arm/Group | IPL / Tri-Luma® Cream and IPL / Inactive Control Cream
Started | 56
Completed | 52
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Final visit 40 days out of window | 1

BASELINE CHARACTERISTICS:
Arm/Group | IPL / Tri-Luma® Cream and IPL / Inactive Control Cream
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were a Success or Failure With Regards to Melasma Severity at Week 10 as Evaluated Using the Investigator's Global Assessment (IGA) of Melasma
Description: Number of participants who were a success or failure with regards to melasma severity at Week 10 as evaluated using the Investigator's Global Assessment (IGA) of melasma (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe) with Clear / Almost Clear being success and all others being failure
Time Frame: Baseline to week 10
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Groups:
- Intense Pulsed Light (IPL) / Tri-Luma® Cream: Intense Pulsed Light (IPL) /fluocinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05%
- Intense Pulsed Light (IPL) / Inactive Control Cream: Intense Pulsed Light (IPL) / Cetaphil® Moisturizing Cream
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
participants
  Success | 32 | 13
  Failure | 24 | 43
  Missing | 0 | 0

2. Secondary Outcome: Number of Participants Who Were a Success or Failure With Regards to Melasma Severity at Week 6 Using the Investigator's Global Assessment (IGA) of Melasma With Clear/Almost Clear Being Success and All Others Being Failure
Description: Number of participants who were a success or failure with regards to melasma severity at Week 6 as evaluated using the Investigator's Global Assessment (IGA) of melasma (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe) with Clear / Almost Clear being success and all others being failure
Time Frame: Baseline to week 6
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Groups:
- Intense Pulsed Light (IPL) / Tri-Luma® Cream: Intense Pulsed Light (IPL) / fluocinolone acetonide 0.01%, hydroquinone 4%, tretinoin 0.05%
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
participants
  Success | 23 | 8
  Failure | 33 | 48
  Missing | 0 | 0

3. Secondary Outcome: Degree of Pigmentation (Melanin) Using a Mexameter at Weeks 6 and 10
Description: Degree of pigmentation (melanin) using a Mexameter to record units on a scale at Weeks 6 and 10; units on a scale is a number that represents the presence or absence of melanin in the skin on a scale from 0 - 999 units with 0 units representing no melanin and 999 units representing the maximum amount of melanin.
Time Frame: Baseline to Week 6 and Baseline to Week 10
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
units on a scale
  Week 6 | 27.5 (52.64) | 36.7 (49.41)
  Week 10 | 15.1 (41.6) | 26.2 (43.89)

4. Secondary Outcome: Number of Participants Showing Success or Failure in Improvement of Melasma at Week 6 Using the Investigator's Evaluation of Improvement
Description: Number of participants showing success or failure in improvement of melasma at Week 6 using the Investigator's evaluation of improvement (0 = Worse, 1 = No change, 2 = Improved, 3 = Much improved, 4 = Excellent Improvement) with Improved, Much improved and Excellent Improvement defined as success and Worse or No change being defined as failure
Time Frame: Baseline to week 6
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
participants
  Success | 46 | 40
  Failure | 7 | 13
  Missing | 3 | 3

5. Secondary Outcome: Number of Participants Showing Success or Failure in Improvement of Melasma at Week 10 Using the Investigator's Evaluation of Improvement
Description: Number of participants showing success or failure in improvement of melasma at Week 10 using the Investigator's evaluation of improvement (0 = Worse, 1 = No change, 2 = Improved, 3 = Much improved, 4 = Excellent Improvement) with Improved, Much improved and Excellent Improvement defined as success and Worse or No change being defined as failure
Time Frame: Baseline to week 10
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
participants
  Success | 44 | 37
  Failure | 9 | 16
  Missing | 3 | 3

6. Secondary Outcome: Number of Participants Showing Success or Failure in Improvement of Melasma at Week 6 Using the Subject's Evaluation of Improvement
Description: Number of participants showing success or failure in improvement of melasma at Week 6 using the Subject's evaluation of improvement (0 = Worse, 1 = No change, 2 = Improved, 3 = Much improved, 4 = Excellent Improvement) with Improved, Much improved and Excellent Improvement defined as success and Worse or No change being defined as failure
Time Frame: Baseline to week 6
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
participants
  Success | 48 | 33
  Failure | 5 | 20
  Missing | 3 | 3

7. Secondary Outcome: Number of Participants Showing Success or Failure in Improvement of Melasma at Week 10 Using the Subject's Evaluation of Improvement
Description: Number of participants showing success or failure in improvement of melasma at Week 10 using the Subject's evaluation of improvement (0 = Worse, 1 = No change, 2 = Improved, 3 = Much improved, 4 = Excellent Improvement) with Improved, Much improved and Excellent Improvement defined as success and Worse or No change being defined as failure
Time Frame: Baseline to week 10
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
participants
  Success | 48 | 36
  Failure | 5 | 17
  Missing | 3 | 3

8. Secondary Outcome: Number of Participants With Tolerability Assessments Resulting in Adverse Events
Description: Number of participants with Tolerability assessments (erythema, scaling, dryness, stinging/burning, edema, telangiectasis, darkening or melasma spots) resulting in adverse events
Time Frame: Baseline to week 10
Population: Safety
Measure: Number; unit: participants
Arm/Group | Intense Pulsed Light (IPL) / Tri-Luma® Cream | Intense Pulsed Light (IPL) / Inactive Control Cream
Number analyzed (Participants) | 56 | 56
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), if applicable.
Arm/Group | IPL / Tri-Luma® Cream and IPL / Inactive Control Cream
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.